CLINICAL TRIAL: NCT03761602
Title: The Correlation Between Iodine and Selenium Status in Pregnancy and Risk of Thyroid Disease: a Prospective Registry Study
Brief Title: The Correlation Between Iodine and Selenium Status in Pregnancy and Risk of Thyroid Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rongrong Li (Other)
Responsible Party: Sponsor-Investigator, Rongrong Li, Nutrition physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: ISCMS
Record Dates: First submitted 2018-11-20; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Iodine Excess in Pregnancy; Selenium Excess in Pregnancy; Iodine Deficiency in Pregnancy; Selenium Deficiency in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples Without DNA — urine and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Proper selenium and iodine condition: The subjects should have proper dietary intake of selenium and iodine, according to Chinese Dietary Reference Intakes (DRIs) (intake of selenium 65μg/d and iodine 230 μg/d).
  The Serum iodine concentration are 45-92μg/L，and the urinary I/Cr 150-249μg/g Cr.
  The Serum selenium concentrations are 18-40μg/L.
  Interventions: Other: Not applicable (for observational studies)
- Excessive selenium or iodine condition: The subjects have excessive dietary intake of selenium and iodine, usually more than 2 times of DRIs. The Serum iodine concentration are more than 100μg/L，and the urinary I/Cr more than 300μg/g Cr.
  The Serum selenium concentrations are more than 40μg/L.
  Interventions: Other: Not applicable (for observational studies)
- Insufficient selenium or iodine condition: The subjects have insufficient dietary intake of either selenium or iodine, compared with DRIs. The Serum iodine concentration are less than 45μg/L，and the urinary I/Cr less than150μg/g Cr.
  The Serum selenium concentrations are less than 18μg/L.
  Interventions: Other: Not applicable (for observational studies)

INTERVENTIONS:
Other: Not applicable (for observational studies) — This study is an observational study. No intervention will be administered for research purposes.

SUMMARY:
Two hundred and ninety pregnant women with gestational age less than 20 weeks will be recruited in this study. Selenium and iodine conditions, and risk of thyroid disease will be monitored until termination of pregnancy, with pregnancy outcomes recorded.

DETAILED DESCRIPTION:
The study will recruit 290 pregnant women with gestational age less than 20 weeks. Iodine and selenium condition will be evaluated through dietary recall (on base of Chinese food ingredient information) and biochemical examinations (serum iodine concentrations, urinary iodine concentrations, serum selenium concentrations, etc). The nutritional status of iodine and selenium will be monitored and followed up for all the included subjects throughout the pregnancy. The information of thyroid function and level of anti-TPO and anti-TG will be collected. And all the complications (especially thyroid disease) in pregnancy will also be recorded. All pregnant women will be followed up until the termination of pregnancy, with pregnancy outcomes recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical confirmation of being pregnant.
* Being within less than 20 weeks of gestationa.

Exclusion Criteria:

* Being pregnant but over 20 weeks of gestationa.
* Mentally or psychologically unstable.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred and ninety pregnant women with gestational age less than 20 weeks should be recruited in this study and will be followed up throughout the whole pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
risk of thyroid disease | From date of participant inclusion until the date of termination of pregnancy, assessed up to 8 months
  prevalence of thyroid disease (abnormal thyroid function; development of thyroid antibodies)
pregnancy outcomes | From date of participant inclusion until the date of termination of pregnancy, assessed up to 8 months
  prevalence of premature birth, stillbirth and abortion

SECONDARY OUTCOMES:
prevalence of other pregnant complications | From date of participant inclusion until the date of termination of pregnancy, assessed up to 8 months
  prevalence of gestational diabetes mellitus, gestational hypertension, dyslipidemia, etc.
prevalence of thyroid disease in neonates | From date of birth to 4 weeks after birth
  prevalence of thyroid disease (abnormal thyroid function; development of thyroid antibodies，or findings of thyroid nodules) in neonates

IPD SHARING:
Plan to Share IPD: No